CLINICAL TRIAL: NCT06237634
Title: Comparison Of The Effectiveness Of Ultrasound Acrossed Corticosteroid And Ozone Injection In Patıents With Carpal Tunnel Syndrome
Brief Title: Corticosteroid And Ozone Injection In Patıents With Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kayseri City Hospital (Other Government)
Responsible Party: Principal Investigator, Havva Talay Calıs, Prof.Dr., Kayseri City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Kayseri CH
Record Dates: First submitted 2023-08-08; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Carpal Tunnel Syndrome
Keywords: ozone injection; corticosteroid injection; carpal tunnel sendromu; ultrasound guided injection
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Splints; Exercise; Counseling; Ozone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Active Comparator): First group (30 people): A hand-wrist support splint and tendon shifting exercises were applied to the upper extremity of the affected side..
  Interventions: Other: splint and exercise and advices
- corticosteroid group (Active Comparator): Second group (30 people): In addition to the treatment and recommendations given to the first group, 40 mg (1 ml) triamcinolone acetonide was injected into the wrist under ultrasound guidance.
  Interventions: Other: splint and exercise and advices; Other: Triamsinolon Asetonid ozone
- ozone group (Experimental): Third group (30 people): In addition to the treatment and recommendations given to the first group, the affected side was injected with ultrasound-guided 3 cc ozone (O2-O3) into the wrist with a concentration of 10 micrograms/ml.
  Interventions: Other: splint and exercise and advices; Other: ozone

INTERVENTIONS:
Other: splint and exercise and advices — A hand-wrist support splint and tendon shifting exercises were applied to the upper extremity of the affected side.
Other: Triamsinolon Asetonid ozone — 40 mg (1 ml) of triamcinolone acetonide was injected to the median nerve's around at wrist level under ultrasound guidance.
  Arms: corticosteroid group
Other: ozone — In addition to the treatment and recommendations given to the first group, the affected side was injected with ultrasound-guided 3 cc ozone (O2-O3) into the wrist with a concentration of 10 micrograms/ml.
  Arms: ozone group

SUMMARY:
There are a limited number of studies on the use of ozone in CTS.The aim of this clinical study is to compare the effectiveness of corticosteroid injections and ozone injections added to splint and exercise therapy in mild-moderate CTS patients..

106 patients included in the study were randomized and divided into three groups. During the follow-up, a total of 90 patients, 30 patients in each group, completed the study.

DETAILED DESCRIPTION:
106 patients included in the study were randomized and divided into three groups.

During the follow-up, a total of 90 patients, 30 patients in each group, completed the study.

Neutral hand-wrist rest splint and tendon-nerve gliding exercises were given to 30 patients included in the control group.

In addition to the treatment given to the first group, 40 mg (1 ml) triamcinolone acetonide was injected under USG guidance to 30 patients included in the corticosteroid group.

In addition to splint and exercise therapy, 3 cc ozone (O2-O3), 10 micrograms were injected under USG guidance to 30 patients in the ozone group.

Patients in all three groups were evaluated at the beginning of treatment, 6 weeks and 3 months after treatment.

Evaluation methods include provocative tests (Tinnel, Phallen, Flick tests), visual analogue scale (VAS) numbness day/night and VAS pain scores, sensory tests (two-point discrimination and Semmes Weinstein monofilament test (SWMT)), hand and finger grip strengths. measurement, Boston carpal tunnel syndrome questionnaire (BCTA), median nerve cross-sectional area (MSCA) measurement with USG and electrophysiological parameters were used.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-70, male or female.
* Clinically and electrophysiologically diagnosed with mild or moderate CTS
* Having symptoms for 1 month or longer
* No contraindications for corticosteroid and ozone application
* Patients whose consent was obtained to participate in the study

Exclusion Criteria:

* Under 18 years old and over 70 years old
* Having a severe CTS
* Having thenar atrophy
* Those with diabetes, thyroid and kidney disease and CTS developing secondary to this
* Those with previous traumatic nerve injury, peripheral nerve injury or surgery
* Those with a diagnosis of polyneuropathy
* Having rheumatic disease
* With known radiculopathy
* are pregnant
* Known G6PD deficiency, hyperthyroidism, thrombocytopenia, severe cardiovascular instability
* Those who have infection, burns, cuts or skin integrity in the skin area to be treated
* Cognitive disorder, severe psychiatric illness
* Those with diabetes, thyroid and kidney disease and CTS developing secondary to this
* Patients who have not received corticosteroid or ozone injection in the last 3 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-04-10 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Boston Carpal Tunnel Syndrome Questionnaire | at baseline, week 6, week 12
  The BCTQ comprises two subscales. The Symptom Severity Scale yields PRO data on the level of symptoms, while the Functional Status Scale assesses the level of hand function. The Symptom Severity Scale consists of 11 items assessing pain, paresthesia, numbness, weakness, nocturnal symptoms, and difficulty of grasping. The Functional Status Scale contains eight items, which assess functional deficits in the following domains: writing, buttoning clothes, holding a book while reading, gripping a telephone handle, opening jars, performing household chores, carrying grocery bags, bathing and dressing. Each item is scored from 1 (no symptoms/difficulties) to 5 (the worst symptoms/cannot perform the activity at all). The mean score for each scale is calculated, resulting in a score between 1 and 5, with higher scores indicating worse symptoms or function. A Finnish version of the BCTQ, which was used in this study, has been previously validated

SECONDARY OUTCOMES:
VAS | at baseline, week 6, week 12
  Visual analog scale A Visual Analogue Scale (VAS) is one of the pain rating scales used for the first time in 1921 by Hayes and Patterson. It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms. For example, the amount of pain that a patient feels ranges across a continuum from none to an extreme amount of pain.
  Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
ultrasound measurements | at baseline, week 6, week 12
  median nerve diameter measurement
EMG measurements | at baseline, week 6, week 12
  median nerve latancy,amplitud, velocity measurements

CONTACTS AND LOCATIONS:
Overall Officials: HAVVA TALAY CALIS, PROF. DR, Principal Investigator — Kayseri City Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - health sciences university Kayseri medicine faculty, Kayseri
  - Health Sciences University, Kayseri Medicine Faculty, Kayseri City Hospital, Kayseri

IPD SHARING:
Plan to Share IPD: No